CLINICAL TRIAL: NCT00991484
Title: Collagen-subtype Analysis in Subcutaneous Tissue and Genetic Analysis on Patients From Families With a Tendency to Hernias
Brief Title: Collagen Analysis and Genetic Analysis of Families With Tendency to Hernias
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Herlev Hospital (Other)
Responsible Party: Jakob Burcharth, MD., Herlev Hospital, Department of surgical Gastroenterology
Other Study IDs: H-4-2009-123
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Hernia
Keywords: ventral; inguinal; hernia; inheritance; genetics
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples and subcutaneous tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- control group
- individuals from hernia-family

SUMMARY:
Analysis of collagen subtype subcutaneously and genetic analysis of patients from families with a tendency to hernias. Furthermore circulating biomarkers and biomarkers extracted from the subcutaneously tissue such as MMP's (matrix metallo proteinases) and TIMP's (tissue inhibitor of metallo proteinases) will be measured.

DETAILED DESCRIPTION:
Research has shown relationship between hernias and collagen subtype I/III ratio, biomarkers such as MMP's TIMP's and other diseases such as Ehlers-Danlos, Marfans syndrome, AAA (abdominal aortic aneurysms), diverticulosis and rectal prolapse. Furthermore has research raised hypothesis about inheritance of hernias. The investigators are performing genetic examination combined with analysis of collagen and biomarkers on patients belonging to families with tendency to hernias.

Other examinations performed on the patients enrolled in this study:

* Ultrasound (US) examination of the abdominal aorta to discover possible abdominal aortic aneurysms.
* Beightons score to evaluate the degree of joint hypermobility.

ELIGIBILITY:
Inclusion Criteria:

* adults over 18 years
* adults must be members of a family where there are presence of hernias in minimum generation.

Exclusion Criteria:

* infections
* pregnant
* mentally ill patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients in Denmark operated or diagnosed with hernias who are member of a family with tendency to hernias.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-12 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Expression of collagen-genes or other relevant genes by microarray analysis compared with presence of hernia | 1 year

SECONDARY OUTCOMES:
Amount of collagen subtypes measured subcutaneously. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Rosenberg, Prof. MD, Study Director — Herlev Hospital; Jakob Burcharth, MD, Principal Investigator — Herlev Hospital
Locations (1):
- Herlev Hospital, Dk-2730, Herlev, Herlev, Denmark